CLINICAL TRIAL: NCT05736549
Title: Yale Steroid Enhanced Versus Exparel Nerveblock TKA Part 2
Acronym: Yale SEVEN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Department of Anesthesiology Faculty Development Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2000031881_a
Record Dates: First submitted 2023-02-07; First posted 2023-02-21 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Total Knee Replacement; Knee Arthroplasty

STUDY DESIGN:
Intervention Model Description: We will conduct a randomized study based on a randomization table generated by a biostatistician on the day of the surgery by the same investigator who will also prepare the study medication and perform the nerve block procedure. Patients follow up will be performed by investigators blinded to group assignments.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- B-LB in left knee and B-DEX-MPA in right knee (Experimental): Participants in this arm will receive B-LB in their left knee and B-DEX-MPA in their right knee.
  Nerve block with (B-LB): A medication mixture of 40 ml (20 ml LB and 20 ml 0.25% plain bupivacaine) will be prepared, of which 20 ml will be used in Adductor canal block, 10 ml will be used in iPACK block and 5 ml each will be used in medial upper and lateral upper genicular nerve block, respectively.
  Nerve block with (B-DEX-MPA): A medication mixture of 40 ml (40 ml 0.25% plain bupivacaine, 10 mg DEX and 80 mg MPA) will be prepared, of which 20 ml will be used in Adductor canal block, 10 ml will be used in iPACK block and 5 ml each will be used in medial upper and lateral upper genicular nerve block, respectively.
  Interventions: Drug: Bupivacaine-Liposomal Bupivacaine; Drug: Bupivacaine -Dexamethasone Sodium Phosphate-Methylprednisolone Acetate
- B-LB in right knee and B-DEX-MPA in left knee (Experimental): Participants in this arm will receive B-LB in their right knee and B-DEX-MPA in their left knee.
  Nerve block with (B-LB): A medication mixture of 40 ml (20 ml LB and 20 ml 0.25% plain bupivacaine) will be prepared, of which 20 ml will be used in Adductor canal block, 10 ml will be used in iPACK block and 5 ml each will be used in medial upper and lateral upper genicular nerve block, respectively.
  Nerve block with (B-DEX-MPA): A medication mixture of 40 ml (40 ml 0.25% plain bupivacaine, 10 mg DEX and 80 mg MPA) will be prepared, of which 20 ml will be used in Adductor canal block, 10 ml will be used in iPACK block and 5 ml each will be used in medial upper and lateral upper genicular nerve block, respectively.
  Interventions: Drug: Bupivacaine-Liposomal Bupivacaine; Drug: Bupivacaine -Dexamethasone Sodium Phosphate-Methylprednisolone Acetate

INTERVENTIONS:
Drug: Bupivacaine-Liposomal Bupivacaine — A medication mixture of 40 ml (20 ml LB and 20 ml 0.25% plain bupivacaine) will be prepared, of which 20 ml will be used in Adductor canal block, 10 ml will be used in iPACK block and 5 ml each will be used in medial upper and lateral upper genicular nerve block, respectively.
  Other Names: B-LB
Drug: Bupivacaine -Dexamethasone Sodium Phosphate-Methylprednisolone Acetate — A medication mixture of 40 ml (40 ml 0.25% plain bupivacaine, 10 mg DEX and 80 mg MPA) will be prepared, of which 20 ml will be used in Adductor canal block, 10 ml will be used in iPACK block and 5 ml each will be used in medial upper and lateral upper genicular nerve block, respectively.
  Other Names: B-DEX-MPA

SUMMARY:
The objective of this study is to investigate the efficacy of Dexamethasone sodium phosphate plus Methylprednisolone acetate in combination with plain bupivacaine ((B-DEX-MPA) compared with Liposomal Bupivacaine in combination with plain bupivacaine (B-LB) on post-surgical pain control among patients undergoing bilateral total knee arthroplasty (TKA) to asses if perineural B-DEX-MPA will result in superior analgesia efficacy as compared to B-LB.

This study will also assess if perineural B-DEX-MPA results in improved quality of postoperative recovery as compared to B-LB.

DETAILED DESCRIPTION:
This phase 2 clinical trial will investigate the efficacy of Dexamethasone sodium phosphate (DEX) plus Methylprednisolone acetate (MPA) in combination with plain bupivacaine (B) compared with Liposomal Bupivacaine (LB) in combination with plain bupivacaine on post-surgical pain control among patients undergoing bilateral total knee arthroplasty (TKA).

The primary objective of this study is to investigate the efficacy of Dexamethasone sodium phosphate (DEX) plus Methylprednisolone acetate (MPA) in combination with plain bupivacaine (B) compared with Liposomal Bupivacaine (LB) in combination with plain bupivacaine on post-surgical pain control among patients undergoing total knee arthroplasty (TKA). The secondary objective of this study is to test the effects of perineural use of B-DEX-MPA vs B-LB on the quality of postoperative recovery as well as surgical outcome and neuropathic pain among patients undergoing bilateral TKA.

This study will also assess if perineural B-DEX-MPA results in improved quality of postoperative recovery as compared to B-LB.

This will be a single center study at Yale New Haven Hospital (YNHH) performed at two clinical sites: York St. Campus (York Street, New Haven) and St. Raphael Campus (Chapel Street, New Haven). An anticipated 66 participants who are scheduled for primary, elective bilateral TKA will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists status I, II and III, elective, primary, bilateral TKA planned for spinal anesthesia with plain 0.5% bupivacaine.

Exclusion Criteria:

* Refusal of consent
* Pregnancy
* Conditions making the patient unable to fill out questionnaire online, through email or over the phone including with cognitive dysfunction, psychiatric disorder, or non-English speaking patients, or lack of internet access which would prevent post discharge follow-up electronically
* Coagulopathy
* Allergy to or for any other reasons cannot use Acetaminophen, Celebrex, local anesthetic bupivacaine, DEX, MPA or LB
* Patients on any amounts of opioids within one month of the surgery date, any substance abuse such as regular marijuana user (more frequent than once per month)
* Insulin dependent or uncontrolled diabetes defined as, day of surgery finger stick glucose >200mg/dl, or HbA1C > 8.0%
* Peripheral Nerve Block site or systemic infection
* Immune compromise (e.g., HIV, chronic glucocorticoid use)
* Severe pre-existing neuropathy
* TKA for indications other than osteoarthritis such as post-traumatic injury or rheumatoid arthritis, history of surgery in the ipsilateral knee joint, revision TKA or bilateral TKA
* Severe hepatic or renal dysfunction (GFR <50 ml/min)
* Actual body weight <60 kg
* Patients with active or latent peptic ulcers, diverticulitis, fresh intestinal anastomoses, and non-specific ulcerative colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change in Postoperative Knee Pain Score | Day 1 and Day 2
  Average postoperative knee pain scores for the first two postoperative days using Visual analogue scale (VAS) pain score. Score range from 0 (no pain) to 10 (worst pain possible).
Postoperative opioid consumption | From anesthesia end time to discharge time, up to 48 hours
  In-hospital postoperative opioid consumption in oral milligram morphine equivalent (OME) will be monitored up to 48-hour between anesthesia end time and discharge time

SECONDARY OUTCOMES:
Average Postoperative Knee Pain Score | Day 7
  Average postoperative knee pain scores for each surgical knee for postoperative day 7 using Visual analogue scale (VAS) pain score. Score range from 0 (no pain) to 10 (worst pain possible).
Worst and best pain score | Day 1, Day 2 and Day 7
  Worst and best postoperative knee pain scores for each surgical knee for days 1, 2 and 7 using Visual analogue scale (VAS) pain score. Score range from 0 (no pain) to 10 (worst pain possible).
Change in functional pain using Brief Pain Inventory (BPI) | baseline, 6 weeks and 3 months
  Compare functional pain using the BPI at baseline, 6 weeks and 3 months. The BPI scale defines pain as follows: Score: 1 - 4 = Mild Pain, Score: 5 - 6 = Moderate Pain, Score: 7 - 10 = Severe Pain.
Change in neuropathic pain using PainDetect | baseline, 6 weeks and 3 months
  Compare neuropathic pain at baseline, 6 weeks and 3 months using PainDetect: a nine-item questionnaire that consists of seven sensory symptom items for pain that are graded from 0= never to 5= strongly, one temporal item on pain-course pattern graded -1 to +1, and one spatial item on pain radiation graded 0 for no radiation or +2 for radiating pain.
Persistent opioid use using Yale Postoperative Recovery Scale | Day 7, 6 weeks and 3 months
  Persistent opioid use will be compared using the Yale Postoperative Recovery Scale on postoperative day 7, 6 weeks and 3 months. It is comprised of 3 free-text questions: Is patient still taking opioid medications, Yes or No; The number of pills left in pill box;and Has the patient needed a prescription refill, Yes or No.
Persistent opioid use using NarX | 6 weeks and 3 months
  Persistent opioid use will be compared using the NarX score at 6 weeks and 3 months, scores range from 000-999; higher scores indicate more opioid usage
Change in Quality of Recovery 40 questionnaire | Day 1, 2 and 7
  40 questions assessing quality of recovery graded on a five-point Likert scale, total score range from 40 (extremely poor recovery) to 200 (excellent recovery)
Prosthetic joint range of motion | baseline, day 0, day 1 and day 2
  Compare prosthetic joint range of motion for each surgical knee using the patient's electronic medical record as reported by the physical therapist at baseline, day 0, day 1, and day 2
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Global-10 | 6 weeks and 3 months
  The PROMIS Global-10 is a 10-item patient-reported questionnaire that measures changes in general health in which the response options are presented as 5-point scale, 5 (without any difficulty) to 1 (Unable to do). Higher scores indicate a healthier patient.
Change in knee functional status using Knee injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS JR) | 6 weeks and 3 months
  Compare knee functional status using KOOS JR at 6 weeks and 3 months after surgery, Scores range from 0 to 100 with a score of 0 indicating total knee disability and 100 indicating perfect knee health.
Length of stay | from the start of the surgery to discharge from hospital, up to 48 hours
  The patient's post surgical length of stay in the hospital will be compared between treatment groups.
Change in glucose | baseline, day 0, day 1 and day 2
  Compare the change in postoperative serum glucose from baseline.
Change in white blood cell count (WBC) | baseline, day 0, day 1 and day 2
  Compare the change in postoperative WBC from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jinlei Li, MD PhD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale New Haven Hospital Saint Raphael Campus, New Haven, Connecticut
  - Yale New Haven Hospital York Street Campus, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No